CLINICAL TRIAL: NCT06207695
Title: A Brief Group Psychosocial Intervention for Earthquake Survivors: Kahramanmaras Earthquakes
Brief Title: Intervention for Earthquake Survivors
Acronym: BriefGroup
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Cennet Yastıbaş, Clinical Psychologist, PhD, Dokuz Eylul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2023-12-18; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Earthquake
Keywords: earthquake; group intervention; psychological distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brief Psychosocial Intervention (Experimental): The group was leaded by two psychologists trained on trauma and disaster psychology, and group intervention. Each groups lasted 2.50 hours.
  Interventions: Behavioral: Brief Group Intervention

INTERVENTIONS:
Behavioral: Brief Group Intervention — This brief intervention consisted of four sessions. The contents of sessions were psychoeducation, emotion processing, practicing emotion regulation strategies, cognitive processing, reframing thoughts, practicing mindful exercises, strength social support networks, and problem management skills.

SUMMARY:
This program for adults in need of psychological support in earthquake stricken area, Kahramanmaraş, consisted of a brief four-session group psychosocial support intervention. The aim of the project was to test the effectiveness of the intervention program. Intervention program was developed by the psychotherapists, a clinical psychologist holding a PhD degree and a psychiatrist. The general theme was about the strengthening of the personal resources including both external and internal resources. The content of the intervention program is based on the relevant literature.

DETAILED DESCRIPTION:
The 6th of February 2023 earthquakes directly affected 11 provinces of our country and were caused thousands loss of life. Trauma in individuals directly affected by the earthquake Post-Traumatic Stress Disorder, depression, anxiety and various psychological problems. These serious psychological problems affect people's functionality significantly and make daily life more difficult. According to the literature, it is seen that various psychosocial support program for earthquake survivors were applied to improve psychological well-being. The results of these interventions demonstrated the psychosocial interventions were effective to diminish psychological distress. Various organisations and communities have continued to provide psychosocial supports peculiar to the needs of individuals living in earthquake stricken areas for the past eight months after the 6th of February 2023 earthquakes. However, the size of the disaster area and the number of people affected is quite high. Thus, a culturally appropriate group of psychosocial intervention program is needed. In this context, the existing research aiming to reduce psychological distress and improve quality of life in the disaster area were examined by the researchers. A brief psychosocial group intervention was developed. This group intervention aiming to strength resources of individuals consisted of four sessions including psychoeducation of the effects of earthquakes, practicing emotion regulation strategies, mindful techniques. The researchers aimed to test the efficacy of this brief psychosocial group intervention. The researchers used a number of measurement tools including psychological distress, quality of life and resilience.

ELIGIBILITY:
Inclusion Criteria:

* Experienced the 6th of February Earthquake in Kahramanmaraş
* Being literate or above
* Being volunteer to participate in group intervention

Exclusion Criteria:

* Having any current psychological treatment related to earthquake
* Being illiteracy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in psychological distress | Baseline measurement before the intervention begin (pre-intervention), immediately after the completion of the intervention (post-intervention)
  The Turkish version of General Health Scale 12. Higher scores refer worse psychological distress
Change in Affect | Baseline measurement before the intervention begin (pre-intervention), immediately after the completion of the intervention (post-intervention)
  The Turkish version of Positive and Negative Affect Scale. It consists of positive and negative affect.Higher scores of each subscales refer higher level of each of them
Change in Quality of Life | Baseline measurement before the intervention begin (pre-intervention), immediately after the completion of the intervention (post-intervention)
  The Turkish version of Short Form-12 will be used. It consisted of 12 items. Higher scores refer higher quality of life.
Change in Self-Efficacy. | Baseline measurement before the intervention begin (pre-intervention), immediately after the completion of the intervention (post-intervention)
  The Turkish Form of Coping Self-Efficacy (tailored earthtquake) will be used. Higher scores are a clear sign of higher coping self-efficacy.
Change in Resilience | Baseline measurement before the intervention begin (pre-intervention), immediately after the completion of the intervention (post-intervention)
  The Turkish form of resilience will be used. Higher scores refer higher resilience scores.
Change in anxiety | Baseline measurement before the intervention begin (pre-intervention), immediately after the completion of the intervention (post-intervention)
  The Turkish version of Generalized Anxiety Disorder-7 will be used. Higher scores refer higher anxiety
Change in depression | Baseline measurement before the intervention begin (pre-intervention), immediately after the completion of the intervention (post-intervention)
  The Turkish Form of Patient Health Questionnaire. It contains 9 item referring depressive symptoms. High scores are a clear sign of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Cennet Yastıbaş Kaçar, PhD, Study Director — Adana Alparslan Turkes Science and Technology University
Locations (1):
- Kahramanmaraş, Kahramanmaraş, Turkey (Türkiye)